CLINICAL TRIAL: NCT02470624
Title: Chinese Acute Ischemic Stroke Treatment Outcome Registry
Acronym: CASTOR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University First Hospital (Other)
Collaborators: Techpool Bio-Pharma Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Yining Huang, Professor, Peking University First Hospital
Other Study IDs: Neurology-stroke
Record Dates: First submitted 2015-06-10; First posted 2015-06-12 (Estimated); Last update posted 2015-10-23 (Estimated); Status verified 2015-10

CONDITIONS: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Months
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- treatment following current guideline
  Interventions: Other: treatment following current guideline

INTERVENTIONS:
Other: treatment following current guideline

SUMMARY:
This is a multi-center registry study. The investigators will include 10,000 patients with confirmed acute ischemic stroke in China. The aim of the study is to survey current treatment situation in China and compare the effectiveness and safety between different intervention regimens.

DETAILED DESCRIPTION:
Stroke is a common disease in China. Compared to western countries, there are many treatment regimens used in clinical practice in China. But their treatment effects are not well validated. The aim of the study is to survey current treatment situation in China and compare the effectiveness and safety between different intervention regimens.

ELIGIBILITY:
Inclusion Criteria:

1. age ≥18 yesrs
2. confirmed diagnosis of an ischemic stroke
3. admission within 1 week after onset of stroke or within treatment time window for patients of thrombolysis treatment
4. signed informed consent

Exclusion Criteria:

1. with intracerebral hemorrhage
2. with severe morbid (estimated survival duration less than 3 months)
3. could not provide follow-up information

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: acute ischemic stroke patients
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2015-05; Primary Completion 2017-03 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
death or severe disability | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Yining Huang, MD, Principal Investigator — Peking University First Hospital
Locations (1):
- Peking University First Hospital, Beijing, China

REFERENCES:
- [Derived] Huang D, Lu Y, Sun W, Sun W, Sun Y, Huang Y, Song Y, Tai L, Li G, Chen H, Zhang G, Zhang L, Sun X, Qiu J, Wei Y, Jin H. Functional Outcomes of Human Urinary Kallindinogenases in Treatment of Acute Ischemic Stroke. Stroke. 2026 Jan;57(1):63-76. doi: 10.1161/STROKEAHA.124.050188. Epub 2025 Sep 29. PMID 41017461
- [Derived] Lu Y, Sun W, Huang Y, Wang Z, Shen Z, Sun W, Liu R, Li F, Shu J, Peng Q, Jia J, Sun P, Song Y, Jin H; CASTOR Investigators. Comparison of Factors Affecting Quality of Life in Patients with Acute Ischemic Stroke Across Different Stroke Severities. Neurol Ther. 2025 Jun;14(3):1023-1038. doi: 10.1007/s40120-025-00743-9. Epub 2025 Apr 29. PMID 40301282
- [Derived] Wang L, Guan X, Zhou J, Hu H, Liu W, Wei Q, Huang Y, Sun W, Jin X, Li H. Measuring the health outcomes of Chinese ischemic stroke patients based on the data from a longitudinal multi-center study. Qual Life Res. 2025 Jul;34(7):1967-1977. doi: 10.1007/s11136-025-03957-4. Epub 2025 Mar 27. PMID 40146503
- [Derived] Lu Y, Sun P, Jin H, Wang Z, Shen Z, Sun W, Sun Y, Liu R, Li F, Shu J, Qiu Z, Lu Z, Sun W, Zhu S, Huang Y; CASTOR Investigators. Prolonged Hospital Length of Stay Does Not Improve Functional Outcome in Acute Ischemic Stroke. Neurol Ther. 2025 Apr;14(2):593-607. doi: 10.1007/s40120-025-00712-2. Epub 2025 Feb 18. PMID 39964661
- [Derived] Li Y, Ou Q, Lu Y, Shen Z, Li J, Zhang Z, Tai L, Li G, Chen H, Zhang G, Zhang L, Sun X, Qiu J, Wei Y, Zhu S, Wang Z, Sun W, Huang Y. Geographic differences in pharmacotherapy patterns and outcomes of acute ischemic stroke in China. BMC Neurol. 2024 Feb 15;24(1):64. doi: 10.1186/s12883-024-03564-9. PMID 38360588
- [Derived] Sun W, Ou Q, Zhang Z, Qu J, Huang Y. Chinese acute ischemic stroke treatment outcome registry (CASTOR): protocol for a prospective registry study on patterns of real-world treatment of acute ischemic stroke in China. BMC Complement Altern Med. 2017 Jul 6;17(1):357. doi: 10.1186/s12906-017-1863-4. PMID 28683732